CLINICAL TRIAL: NCT02146573
Title: Pediatric Continuity Care Intensivist: Role Implementation and Randomized Control Trial
Brief Title: Pediatric Continuity Care Intensivist
Acronym: CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 14-010987
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Critical Illness
Keywords: Intensive Care Units, Pediatric; Communication; Health personnel; Decision making; Critical Care; Length of Stay; Iatrogenic Disease
MeSH Terms: conditions — Critical Illness; Communication; Iatrogenic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCI Provider for Parent-patient dyad (Experimental): Parents and patients are randomly assigned to a Continuity Care Intensivist (CCI) Provider who has received specialized communication training. The parent-patient dyad will receive standardized care from the CCI throughout their time in the PICU in addition to being assigned a rotating physician of record.
  Interventions: Behavioral: Continuity Care Intensivist Communication Training; Behavioral: Continuity Care Intensivist (CCI) Provider Program
- Usual Care for Parent-patient dyad (No Intervention): Patients and parents randomly assigned to usual care in the PICU which includes the rotation of the physician of record approximately every 7 days. There is no standardized process by which patients may be assigned a primary attending who would follow them throughout their stay. In the usual care arm it may never happen that they are assigned a primary intensivist, regardless of the length of their hospitalization.

INTERVENTIONS:
Behavioral: Continuity Care Intensivist Communication Training — Physicians enrolled in the intervention arm will complete a two to three part communication training. Survey measures of communication competency and burnout will be administered at baseline, after training, and at the end of the study. After the communication training, physicians will undergo an OSCE assessment with a simulated patient to evaluate communication skills. At the end of the study, CCI providers will receive surveys that assess the experience and challenges of the role, repeat surveys assessing competency with communication and frequency of engaging families in goals of care conversations, in addition to a follow-up focus group that will assess their experience with the intervention, the time required and the potential tradeoffs in other duties required by them to participate as a CCI.
  Other Names: CCI Communication Training
  Arms: CCI Provider for Parent-patient dyad
Behavioral: Continuity Care Intensivist (CCI) Provider Program — After undergoing CCI training, CCI providers will fulfill a standardized role with parent-patient dyads:
  * CCI will meet with families on a regular basis and at change of physician of record throughout their entire PICU hospitalization.
  * Help patients/families navigate decisions in concert with preferences and beliefs
  * Help patients/families and other care providers look at "bigger picture"; trajectory of illness, goals, and hopes for the patient.
  * Serve as point person for active intensivists on service and other specialists
  * Help resolve conflict when multiple providers have different opinions on course of action
  Other Names: CCI Provider
  Arms: CCI Provider for Parent-patient dyad

SUMMARY:
This study will implement and evaluate the effects of a pediatric continuity care intensivist program. This study will determine the impact of an additional pediatric intensive care unit (PICU) intensivist on outcomes at the patient and family level. It will also evaluate the training program to prepare the continuity care intensivist (CCI).

DETAILED DESCRIPTION:
This randomized controlled trial will implement and evaluate the effects of a pediatric continuity care intensivist (CCI) program. The study will evaluate how effective the modified communication training for providers is to perform this new role. The primary outcome for the study is whether a CCI will affect several patient level outcomes for patients who have been admitted to the PICU longer than 7 days. Patient length of stay, hospital acquired conditions, time to limitations of interventions and new medical technology will be assessed comparing the intervention and usual care arms. The study will also determine the impact of the CCI program on parent/family satisfaction with provider communication and decision-making for their child.

ELIGIBILITY:
Inclusion Criteria:

CCI Provider

1. Pediatric Intensive Care Unit Attending Physician who volunteers to serve in the role of CCI.

Usual Care (UC) Provider

1. Any Pediatric Intensive Care Unit Attending Physician who is not enrolled as a CCI.

Parent-Patient Dyads

1. Parent/guardian of a child who has been admitted to the Children's Hospital of Philadelphia (CHOP) PICU for ≥7 days after onset of the study
2. Parent/guardian ≥ 18 years old
3. Parent/guardian is English-speaking
4. Child <18 years old at time of enrollment
5. Child has been admitted to the PICU at CHOP for ≥7 days
6. Medical team believed that patient will remain in the PICU for at least another seven days

Exclusion Criteria:

CCI Provider

1. Any medical care provider who is not an attending physician (e.g., Pediatric critical care residents, nurses, and fellows)

UC Provider

1. Any medical care provider who is not an attending physician (e.g., Pediatric critical care residents, nurses, and fellows)
2. Attending physician who is enrolled in the study as a CCI

Parent-Patient Dyads

1. Parent or guardian who has previously participated in the CCI study in a previous hospitalization (in either usual care or intervention arm)
2. Parent or guardian of a child who has already been hospitalized in the PICU >7 days at the onset of the study.
3. Child ≥18 years of age at time of enrollment
4. Child has previously participated in the CCI study in a previous PICU stay (in either usual care or intervention arm)
5. Child has been hospitalized in the PICU >7 days at the onset of the study
6. Child already has a "primary" attending
7. Child has a sibling that has already been enrolled in the study. This child will be ineligible for the study but will be assigned to the same care as the child who is or was enrolled in the study.
8. If contact was not established for enrollment by 14 days after admission, then the patient was no longer considered eligible for enrollment to maintain comparability of length of stay at enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Difference in patient length of stay in the PICU between usual care and intervention arm | up to 600 days
  Length of stay as measured by the Virtual PICU system (VPS) in the PICU.

SECONDARY OUTCOMES:
Difference in number of new technological dependence patients acquire during hospitalization between usual care and intervention arms | up to 600 days
  We will measure new technology dependence like tracheostomy, gastrostomy tube, long term ventilation, bipap using VPS during the PICU hospitalization.
Difference in patient hospital-acquired conditions between usual care and intervention arm | up to 600 days
  Using VPS, investigators will track hospital acquired infections like catheter associated urinary tract infections and ventilator associated pneumonias
Difference in patient length of time on sedation medicines between usual care and intervention arm | up to 600 days
  Investigators will track the length of time on sedation medications used during intubations and when there is other medical equipment like chest tubes that it is not safe for patients to be moving. These medications include midazolam and fentanyl among others.
Difference in patients' new or progressive multiple organ dysfunction syndrome between usual care and intervention arm | up to 600 days
  Investigators will use the VPS designation of multiple organ dysfunction syndrome to characterize system failures like respiratory, renal, cardiac failure.
Difference in patient organ failure free days between usual care and intervention arm | up to 600 days
  Investigators will use the VPS designation of organ failure for systems like renal, respiratory and cardiac.
Difference in patient ventilator free days between usual care and intervention arm | up to 600 days
  Investigators will use the VPS designation for days up to 90 that the patient remains off of mechanical ventilation.
Difference in change in parent preferences for shared decision-making from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  A decision-analysis method will be used to administer and measure parental preferences for shared decision-making. Validation of the measure is completed but not yet published by the principal investigator.
Difference in change in parent preferences for control in decision-making from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  The Control Preferences Scale for Pediatrics (CPS-P), a validated tool, will be used to measure parent's preferences for control in decision-making.
Affects of Parent attachment style on communication preferences | baseline
  The Relationship Questionnaire, a validated measure, will be used to measure parent relationship style, which is based on attachment theory.
Difference in change in parental levels of anxiety and depression from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  Parental levels of hospital anxiety and depression will be measured using the Hospital Anxiety and Depression scale (HADS).
Difference in change in parental levels of positive and negative affect from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  Parental levels of positive and negative affect will be measured using the Positive and Negative Affect Scale (PANAS), a validated tool.
Difference in change in parental levels of anger from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  Parent levels of anger will be measured using PROMIS bank v1.1- Anger scale.
Difference in change in parental levels of hope from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  Parental levels of hope will be measured using the Hope Scale, a validated tool.
Difference in change in Parent/family satisfaction with decision-making from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  Parent satisfaction with decision-making will measured through several question items designed to assess parent satisfaction with making decisions during their child's PICU visit. This measure was developed through extensive literature review and has been evaluated for face validity through cognitive interviewing and pilot testing with parents and families of children admitted to the ICU.
Difference in parent/family satisfaction with communication with their child's PICU physicians between usual care and intervention arm | up to 600 days
  The Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU), a validated tool, will be used to measure parent satisfaction with communication with their child's PICU physician.
Difference in change in parent self-report of medical communication competence from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  The Medical Communication Competence Scale, a partially validated tool, will be used to measure parent self-reported competency with communication.
Difference in change in parent assessment of physician communication competency from baseline to patient discharge between usual care and intervention arm | baseline, up to 600 days
  The Communication Assessment Tool (CAT), a validated tool, will be used to measure parent perceptions of physician competence in interpersonal and communication skills.
Comparison of physician burnout between intervention and control group from baseline up to 600 days | baseline, up to 600 days
  The Maslach Stress and Burnout Inventory, a validated tool, will be used to measure the three aspects of the burnout syndrome: emotional exhaustion, depersonalization, and lack of personal accomplishment.
Physician satisfaction with the communication training and with the CCI experience. | up to 600 days
  Questions written for this study that have been written and piloted will assess the physicians' satisfaction and perceived usefulness of the communication training.
Evaluation of CCI provider experience in role of CCI and its feasibility of larger implementation | up to 600 days
  Both open ended survey questions and focus groups will be qualitatively analyzed to determine the benefits and burdens for providers of serving in the CCI role.
Comparison of physician comfort with end-of-life communication between intervention and control group from baseline up to 600 days | baseline, up to 600 days
  Physician comfort with end-of-life communication will be measured through several question items developed to assess how physicians feel about engaging in end of life discussions. The measure was developed through extensive literature review and has been evaluated for face validity through cognitive interviewing and pilot testing with PICU physicians.
Difference in timing of patient's limitations of interventions to death between usual care and intervention arm | up to 600 days
  As measured by a chart review of timing of limitations of interventions including do not resuscitate (DNR)/ do not intubate (DNI) and other limitations like no escalation of care will be described and the time to event of death will be compared.
Frequency of palliative care consultation between usual care and intervention arm | up to 600 days
  Medical chart review to determine request for and consultation performed by Pediatric Advanced Care Team (palliative care consultation service) will be measured and compared.
Physician competency in communication with families via objective structured clinical examination (OSCE) evaluation | up to 600 days
  CCI providers will be evaluated using a simulated patient and scored using a validated tool for communication skills including empathy in an encounter in the end-of-life setting.
Comparison of physician self-reported communication competency between intervention and control group | baseline, up to 600 days
  The Medical Communication Competence Scale, a partially validated measure will be used to assess physician self-reported competency.
Correlation between amount of CCI contact and parent and patient level outcomes | baseline, up to 600 days
  Investigators will categorize the extent of CCI contact and then determine if there is a correlation between amount of contact and parent and patient level outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Walter, MD, PhD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Board R, Ryan-Wenger N. Long-term effects of pediatric intensive care unit hospitalization on families with young children. Heart Lung. 2002 Jan-Feb;31(1):53-66. doi: 10.1067/mhl.2002.121246. PMID 11805751
- [Background] Balluffi A, Kassam-Adams N, Kazak A, Tucker M, Dominguez T, Helfaer M. Traumatic stress in parents of children admitted to the pediatric intensive care unit. Pediatr Crit Care Med. 2004 Nov;5(6):547-53. doi: 10.1097/01.PCC.0000137354.19807.44. PMID 15530191
- [Background] Needle JS, O'Riordan M, Smith PG. Parental anxiety and medical comprehension within 24 hrs of a child's admission to the pediatric intensive care unit*. Pediatr Crit Care Med. 2009 Nov;10(6):668-74; quiz 674. doi: 10.1097/PCC.0b013e3181a706c9. PMID 19451843
- [Background] Pochard F, Darmon M, Fassier T, Bollaert PE, Cheval C, Coloigner M, Merouani A, Moulront S, Pigne E, Pingat J, Zahar JR, Schlemmer B, Azoulay E; French FAMIREA study group. Symptoms of anxiety and depression in family members of intensive care unit patients before discharge or death. A prospective multicenter study. J Crit Care. 2005 Mar;20(1):90-6. doi: 10.1016/j.jcrc.2004.11.004. PMID 16015522
- [Background] Fauman KR, Pituch KJ, Han YY, Niedner MF, Reske J, LeVine AM. Predictors of depressive symptoms in parents of chronically ill children admitted to the pediatric intensive care unit. Am J Hosp Palliat Care. 2011 Dec;28(8):556-63. doi: 10.1177/1049909111403465. Epub 2011 Mar 30. PMID 21454321
- [Background] Nuss SL, Hinds PS, LaFond DA. Collaborative clinical research on end-of-life care in pediatric oncology. Semin Oncol Nurs. 2005 May;21(2):125-34; discussion 134-44. doi: 10.1016/j.soncn.2004.12.011. PMID 15991662
- [Background] Diaz-Caneja A, Gledhill J, Weaver T, Nadel S, Garralda E. A child's admission to hospital: a qualitative study examining the experiences of parents. Intensive Care Med. 2005 Sep;31(9):1248-54. doi: 10.1007/s00134-005-2728-8. Epub 2005 Jul 15. PMID 16021417
- [Background] Colville G, Darkins J, Hesketh J, Bennett V, Alcock J, Noyes J. The impact on parents of a child's admission to intensive care: integration of qualitative findings from a cross-sectional study. Intensive Crit Care Nurs. 2009 Apr;25(2):72-9. doi: 10.1016/j.iccn.2008.10.002. Epub 2008 Nov 18. PMID 19019677
- [Background] Back AL, Arnold RM, Baile WF, Fryer-Edwards KA, Alexander SC, Barley GE, Gooley TA, Tulsky JA. Efficacy of communication skills training for giving bad news and discussing transitions to palliative care. Arch Intern Med. 2007 Mar 12;167(5):453-60. doi: 10.1001/archinte.167.5.453. PMID 17353492
- [Background] Davidson JE, Powers K, Hedayat KM, Tieszen M, Kon AA, Shepard E, Spuhler V, Todres ID, Levy M, Barr J, Ghandi R, Hirsch G, Armstrong D; American College of Critical Care Medicine Task Force 2004-2005, Society of Critical Care Medicine. Clinical practice guidelines for support of the family in the patient-centered intensive care unit: American College of Critical Care Medicine Task Force 2004-2005. Crit Care Med. 2007 Feb;35(2):605-22. doi: 10.1097/01.CCM.0000254067.14607.EB. PMID 17205007
- [Background] Namachivayam P, Shann F, Shekerdemian L, Taylor A, van Sloten I, Delzoppo C, Daffey C, Butt W. Three decades of pediatric intensive care: Who was admitted, what happened in intensive care, and what happened afterward. Pediatr Crit Care Med. 2010 Sep;11(5):549-55. doi: 10.1097/PCC.0b013e3181ce7427. PMID 20124947
- [Background] Feudtner C, Christakis DA, Connell FA. Pediatric deaths attributable to complex chronic conditions: a population-based study of Washington State, 1980-1997. Pediatrics. 2000 Jul;106(1 Pt 2):205-9. PMID 10888693
- [Background] Azoulay E, Pochard F, Chevret S, Lemaire F, Mokhtari M, Le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Meeting the needs of intensive care unit patient families: a multicenter study. Am J Respir Crit Care Med. 2001 Jan;163(1):135-9. doi: 10.1164/ajrccm.163.1.2005117. PMID 11208638
- [Background] Johnson D, Wilson M, Cavanaugh B, Bryden C, Gudmundson D, Moodley O. Measuring the ability to meet family needs in an intensive care unit. Crit Care Med. 1998 Feb;26(2):266-71. doi: 10.1097/00003246-199802000-00023. PMID 9468163
- [Background] Curtis JR, Ciechanowski PS, Downey L, Gold J, Nielsen EL, Shannon SE, Treece PD, Young JP, Engelberg RA. Development and evaluation of an interprofessional communication intervention to improve family outcomes in the ICU. Contemp Clin Trials. 2012 Nov;33(6):1245-54. doi: 10.1016/j.cct.2012.06.010. Epub 2012 Jul 6. PMID 22772089
- [Background] Schneiderman LJ. Ethics consultation in the intensive care unit. Curr Opin Crit Care. 2005 Dec;11(6):600-4. doi: 10.1097/01.ccx.0000179933.54508.7a. PMID 16292067
- [Background] Schneiderman LJ. Effect of ethics consultations in the intensive care unit. Crit Care Med. 2006 Nov;34(11 Suppl):S359-63. doi: 10.1097/01.CCM.0000237078.54456.33. PMID 17057599
- [Background] Schneiderman LJ, Gilmer T, Teetzel HD. Impact of ethics consultations in the intensive care setting: a randomized, controlled trial. Crit Care Med. 2000 Dec;28(12):3920-4. doi: 10.1097/00003246-200012000-00033. PMID 11153636
- [Background] Schneiderman LJ, Gilmer T, Teetzel HD, Dugan DO, Blustein J, Cranford R, Briggs KB, Komatsu GI, Goodman-Crews P, Cohn F, Young EW. Effect of ethics consultations on nonbeneficial life-sustaining treatments in the intensive care setting: a randomized controlled trial. JAMA. 2003 Sep 3;290(9):1166-72. doi: 10.1001/jama.290.9.1166. PMID 12952998
- [Background] Gilmer T, Schneiderman LJ, Teetzel H, Blustein J, Briggs K, Cohn F, Cranford R, Dugan D, Kamatsu G, Young E. The costs of nonbeneficial treatment in the intensive care setting. Health Aff (Millwood). 2005 Jul-Aug;24(4):961-71. doi: 10.1377/hlthaff.24.4.961. PMID 16136635
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Contro N, Larson J, Scofield S, Sourkes B, Cohen H. Family perspectives on the quality of pediatric palliative care. Arch Pediatr Adolesc Med. 2002 Jan;156(1):14-9. doi: 10.1001/archpedi.156.1.14. PMID 11772185
- [Background] Leach MJ. Rapport: a key to treatment success. Complement Ther Clin Pract. 2005 Nov;11(4):262-5. doi: 10.1016/j.ctcp.2005.05.005. Epub 2005 Jun 28. PMID 16290897
- [Background] Kimberlin C, Brushwood D, Allen W, Radson E, Wilson D. Cancer patient and caregiver experiences: communication and pain management issues. J Pain Symptom Manage. 2004 Dec;28(6):566-78. doi: 10.1016/j.jpainsymman.2004.03.005. PMID 15589081
- [Background] DeLemos D, Chen M, Romer A, Brydon K, Kastner K, Anthony B, Hoehn KS. Building trust through communication in the intensive care unit: HICCC. Pediatr Crit Care Med. 2010 May;11(3):378-84. doi: 10.1097/PCC.0b013e3181b8088b. PMID 19770787
- [Background] Meert KL, Eggly S, Pollack M, Anand KJ, Zimmerman J, Carcillo J, Newth CJ, Dean JM, Willson DF, Nicholson C; National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Parents' perspectives on physician-parent communication near the time of a child's death in the pediatric intensive care unit. Pediatr Crit Care Med. 2008 Jan;9(1):2-7. doi: 10.1097/01.PCC.0000298644.13882.88. PMID 18477906
- [Background] Heyland DK, Rocker GM, Dodek PM, Kutsogiannis DJ, Konopad E, Cook DJ, Peters S, Tranmer JE, O'Callaghan CJ. Family satisfaction with care in the intensive care unit: results of a multiple center study. Crit Care Med. 2002 Jul;30(7):1413-8. doi: 10.1097/00003246-200207000-00002. PMID 12130954
- [Background] Mack JW, Wolfe J, Cook EF, Grier HE, Cleary PD, Weeks JC. Hope and prognostic disclosure. J Clin Oncol. 2007 Dec 10;25(35):5636-42. doi: 10.1200/JCO.2007.12.6110. PMID 18065734
- [Background] Epstein D, Unger JB, Ornelas B, Chang JC, Markovitz BP, Moromisato DY, Dodek PM, Heyland DK, Gold JI. Psychometric evaluation of a modified version of the family satisfaction in the ICU survey in parents/caregivers of critically ill children*. Pediatr Crit Care Med. 2013 Oct;14(8):e350-6. doi: 10.1097/PCC.0b013e3182917705. PMID 23863815
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Pyke-Grimm KA, Degner L, Small A, Mueller B. Preferences for participation in treatment decision making and information needs of parents of children with cancer: a pilot study. J Pediatr Oncol Nurs. 1999 Jan;16(1):13-24. doi: 10.1177/104345429901600103. PMID 9989013
- [Background] Cegala DJ, Coleman MT, Turner JW. The development and partial assessment of the medical communication competence scale. Health Commun. 1998;10(3):261-88. doi: 10.1207/s15327027hc1003_5. PMID 16370986
- [Background] Snyder CR, Harris C, Anderson JR, Holleran SA, Irving LM, Sigmon ST, Yoshinobu L, Gibb J, Langelle C, Harney P. The will and the ways: development and validation of an individual-differences measure of hope. J Pers Soc Psychol. 1991 Apr;60(4):570-85. doi: 10.1037//0022-3514.60.4.570. PMID 2037968
- [Background] Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007 Aug;67(3):333-42. doi: 10.1016/j.pec.2007.05.005. Epub 2007 Jun 18. PMID 17574367